CLINICAL TRIAL: NCT05233215
Title: GROW Support (Glioma Specialists Reaching Out With Support): Assessment of a Comprehensive Support Program for Low Grade Glioma Patients Post-treatment
Brief Title: GROW (Glioma Specialists Reaching Out With Support) Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-650
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Low-grade Glioma; Survivorship; Care Giving Burden
Keywords: Low-grade Glioma; Survivorship; Care Giving Burden
MeSH Terms: conditions — Caregiver Burden | interventions — Palliative Care; Allied Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GROW Support Program (Experimental): Patient participants will fill out questionnaires about emotional and physical health with responses used to develop an individualized survivorship plan conducted through 1x monthly virtual or in-clinic check-ins as well as GROW support meetings as needed for 6 months.
  Caregiver participants will fill out questionnaires used to develop patient individualized survivorship plan and participate in 1x monthly check-in meetings with patients or separately for 6 months.
  Interventions: Behavioral: GROW (Glioma Specialists Reaching Out With Support) Support Program

INTERVENTIONS:
Behavioral: GROW (Glioma Specialists Reaching Out With Support) Support Program — Follow-up survivorship care plan for patients and caregivers
  Other Names: Support Program

SUMMARY:
This research study is being done to test a participant and caregiver-driven model of follow-up survivorship care,GROW Support (Glioma Specialists Reaching Out With Support), for post-treatment, low grade glioma patients.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which examines if a supportive intervention for people with low grade gliomas (LGGs) and their caregivers is acceptable and feasible to patients and their caregivers.

The research study procedures include: screening for eligibility and study interventions including filling out questionnaires and virtual or in-clinic supportive follow up visits to identify additional supportive needs that may arise.

Participants will be in this research study for up to 6 months.

It is expected that about 40 people will take part in this research study.

The Levitan-Zabin Fund for GROW Support is supporting this research study by providing funds for research team members to do this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria include:

  * Must be at least 18 years of age;
  * Diagnosed with low grade glioma (WHO grade 1 or 2)
  * Completed active treatment within the last 2 years and are undergoing surveillance follow-up
  * Must have at least one caregiver willing to participate as indicated below
  * Read and comprehend English such that they are able to complete required intervention sessions and psychosocial battery in English and are able to understand and willing to sign an electronic informed consent document.
  * Confirms willingness to undergo initial and follow-up questionnaire battery.
* Caregiver inclusion criteria include:

  * Must be at least 18 years of age
  * Read and comprehend English such that they are able to complete required intervention sessions and psychosocial battery in English and able to understand and willing to sign an electronic informed consent document
  * Consider themselves personally involved in the patient's care and decisions about the care they receive.

Exclusion Criteria:

* Bipolar disorder,
* Psychotic disorders and
* Confusion or altered mental state that would prohibit understanding and giving of informed consent. However, if the patient's bipolar disorder or psychotic disorder is currently treated/managed, the patient will be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Retention Rate | 6 months
  Primary outcome is feasibility as defined by 60% of the eligible participants and their caregivers being recruited into the study and completing the initial assessment and associated survivorship plan

SECONDARY OUTCOMES:
Abbreviated Acceptability Rating Profile | 6 months
  Acceptability of this supportive program ("GROW Support") for patients and their caregivers will be assessed by the Abbreviated Acceptability Rating Profile and based on in-depth semi-structured interview with one of the study investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Sannes, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu